CLINICAL TRIAL: NCT06900374
Title: RF-Vaginale : Randomised Phase III Trial Evaluating the Efficacy and Safety of Vaginal Radiofrequency in the Management of Vulvovaginal Atrophy and Dryness in Patients Treated for Breast Cancer
Brief Title: Efficacy and Safety of Vaginal Radiofrequency for Vulvovaginal Atrophy in Breast Cancer Patients
Acronym: RF-Vaginale
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: MATMATECH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-Vaginale-2401; 2024-A01126-41 (Other: ANSM)
Record Dates: First submitted 2025-02-24; First posted 2025-03-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Vaginal Dryness; Breast Cancer; Vulvovaginal Atrophy
Keywords: Vaginal dryness; vaginal atrophy; vaginal radiofrequency; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The evaluator will be blinded to the intervention (different investigator for vaginal radiofrequency sessions and clinical evaluation consultations) Blinding will be lifted after the 6-month evaluation, with the possibility of radiofrequency treatment for control group patients who are insufficiently relieved
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal radiofrequency treatment (Experimental): The evaluator will be blinded to the intervention (different investigator for vaginal radiofrequency sessions and clinical evaluation consultationsup to 6 months, M0, M3 and M6).
  The blinding will be lifted after the 6-month evaluation, with the possibility of radiofrequency treatment for patients in the control group who are not sufficiently relieved.
  Interventions: Device: GynWave-360; Other: Local hydratation
- Reference treatment (Active Comparator): Local hydration: hyaluronic acid-based treatment, 3 applications per week Possibility of resorting to associated measures chosen by the investigator (physical therapy, vaginal dilators, etc.), excluding physical treatments (vaginal laser, photobiomodulation, PRP injection, hyaluronic acid injection, or lipomodelling).
  Interventions: Other: Local hydratation

INTERVENTIONS:
Device: GynWave-360 — For patients randomized to the experimental group:
  3 sessions of 20 minutes each, spaced 4 to 6 weeks apart (M0, M1, M2) ideally, with +/- 1 maintenance session between 8 and 12 months after the first session (M8-12).
  Arms: Vaginal radiofrequency treatment
Other: Local hydratation — Reference treatment combining local hydration (hyaluronic acid-based treatment, 3 times a week), with the possibility of using associated measures at the investigator's discretion (physiotherapy, vaginal dilators, etc.).

SUMMARY:
This Phase III, randomized, balanced, parallel-group, multicenter trial aims to evaluate the effect of vaginal radiofrequency on symptoms of vaginal dryness at six months. The study compares vaginal radiofrequency treatment with non-hormonal hydration therapy in a population of patients undergoing adjuvant hormonal therapy with aromatase inhibitors, with or without LHRH agonists, for breast cancer.

Patients will be randomly assigned to one of two parallel treatment groups until the six-month assessment:

The first group will receive the reference treatment, which consists of local hydration using a hyaluronic acid-based treatment applied three times a week. Additionally, investigators may incorporate supportive measures at their discretion, such as physiotherapy or vaginal dilators.

The second group will receive the same reference treatment combined with vaginal radiofrequency therapy. This intervention consists of three sessions, each spaced 4 to 6 weeks apart.

DETAILED DESCRIPTION:
This study aims to see if vaginal radiofrequency therapy can help reduce vaginal dryness in women receiving hormone therapy for breast cancer.

The participants are divided into two groups:

One group will use a non-hormonal vaginal moisturizer (hyaluronic acid) three times a week. If needed, they can also use other supportive treatments like physiotherapy or vaginal dilators.

The other group will receive the same moisturizer treatment but will also have three sessions of vaginal radiofrequency therapy, with each session spaced 4 to 6 weeks apart.

After six months, researchers will compare the two groups to see if vaginal radiofrequency provides additional benefits in relieving vaginal dryness.

ELIGIBILITY:
INCLUSION CRITERIA :

* Patient over 40 years
* Presenting disabling vaginal dryness symptoms despite well-administered local moisturizing treatment, attested by a vaginal dryness score ≥3
* Patient undergoing adjuvant treatment for breast cancer
* Patient treated with aromatase inhibitors +/- LHRH agonist for at least 3 months with a planned remaining duration of at least 12 months
* Patient affiliated to a social security organization
* Patient having signed the informed consent for the present study

EXCLUSION CRITERIA:

* Contraindications related to the radiofrequency technique:

  * Ongoing urinary tract infection
  * Pacemaker
  * IUD intrauterine device
  * Pregnancy
* Mucocutaneous disease with vulvovaginal localization: infection, sore, scleratrophic lichen, psoriasis, eczema, etc.
* Neurodegenerative disease with perineal involvement
* Current or recent treatment (within the last 12 months) with other physical methods: vaginal laser, photobiomodulation, PRP injection, hyaluronic acid injection or lipo-modeling.
* Pregnant or breast-feeding women
* Patients under guardianship or trusteeship.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical scale for vaginal dryness according to patient | The main analysis will focus on assessment at 6 months (M6). This endpoint will also be assessed at baseline (M0), 3 and 12 months (M3, M12).
  Patient-rated 0-10 Numerical Rating Scale for vaginal dryness, minimum value =0; maximum value = 10; where 0 = No dryness and 10 = Maximum possible dryness.

SECONDARY OUTCOMES:
Patient-Rated 0-10 numerical scale for dyspareunia | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Patient-rated 0-10 numerical rating scale for dyspareunia, minimum value = 0; maximum value = 10; where 0 = No pain during intercourse and 10 = Maximum possible pain
Vaginal Health Index Score (VHIS) : vaginal elasticity score | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Vaginal elasticity is assessed by a physician observer blinded to the treatment group. It is scored on a 5-point scale:
  1. = None
  2. = Poor
  3. = Fair
  4. = Good
  5. = Excellent
  Higher scores indicate better vaginal elasticity.
Vaginal Health Index Score (VHIS) : vaginal fluid volume score | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Vaginal fluid volume is assessed by a physician observer blinded to the treatment group. It is scored on a 5-point scale:
  1. = None
  2. = Scar amount (vault not entirely covered)
  3. = Superficial amount (vault entirely covered)
  4. = Moderate amount
  5. = Normal amount Higher scores indicate greater fluid volume, which reflects better vaginal hydration.
Vaginal Health Index Score (VHIS) : vaginal pH measurement | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Vaginal pH is measured using a pH test strip applied to the vaginal mucosa by a physician observer. The pH is categorized as follows:
  1. = ≥6.1
  2. = 5.6-6.0
  3. = 5.1-5.5
  4. = 4.7-5.0
  5. = ≤4.6 Lower values indicate a healthier vaginal environment.
Vaginal Health Index Score (VHIS): vaginal epithelial integrity score | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Epithelial integrity is assessed by a physician observer blinded to the treatment group. It is scored on a 5-point scale:
  1. = Petechiae noted before contact
  2. = Bleeds with light contact
  3. = Bleeds with scraping
  4. = Not friable (thin epithelium)
  5. = Normal Higher scores indicate better vaginal epithelial integrity.
Vaginal Health Index Score (VHIS): vaginal moisture score | baseline (M0), 3, 6 and 12 months (M3, M6, M12)
  Vaginal moisture is assessed by a physician observer blinded to the treatment group. It is scored on a 5-point scale:
  1. = None (surface inflamed)
  2. = None (surface non-inflamed)
  3. = Minimal
  4. = Moderate
  5. = Normal Higher scores indicate better vaginal moisture levels.
Side effects of radiofrequency treatment | through study completion: 12 months
  Type of side effects : sensation of heat, redness, erythema, hypersensitivity, dyspareunia, other.
  Time of onset : during the session, immediately after, or more than 24 hours after the session.
  Intensity : graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0), with scores ranging from Grade 1 (mild) to Grade 5 (death). Higher scores indicate greater severity of adverse effects.
  Consequences for the treatment: need to interrupt the session, reduce the radiofrequency temperature, etc.

OTHER OUTCOMES:
Occurrence of discontinuation or modification of hormone therapy | through study completion: 12 months
  - At each follow-up visit 3 months, 6 months, 12 months post-randomization : data collection on any discontinuation of initially prescribed hormone therapy, change of hormone therapy, other changes in treatment, and reasons for these changes.

CONTACTS AND LOCATIONS:
Overall Officials: Julie DEMETZ, MD, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faubion SS, Sood R, Kapoor E. Genitourinary Syndrome of Menopause: Management Strategies for the Clinician. Mayo Clin Proc. 2017 Dec;92(12):1842-1849. doi: 10.1016/j.mayocp.2017.08.019. PMID 29202940
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] Moral E, Delgado JL, Carmona F, Caballero B, Guillan C, Gonzalez PM, Suarez-Almarza J, Velasco-Ortega S, Nieto C; as the writing group of the GENISSE study. Genitourinary syndrome of menopause. Prevalence and quality of life in Spanish postmenopausal women. The GENISSE study. Climacteric. 2018 Apr;21(2):167-173. doi: 10.1080/13697137.2017.1421921. Epub 2018 Feb 7. PMID 29411644
- [Background] Simon JA, Davis SR, Althof SE, Chedraui P, Clayton AH, Kingsberg SA, Nappi RE, Parish SJ, Wolfman W. Sexual well-being after menopause: An International Menopause Society White Paper. Climacteric. 2018 Oct;21(5):415-427. doi: 10.1080/13697137.2018.1482647. Epub 2018 Jul 10. PMID 29987939
- [Background] Nappi RE, Cucinella L, Martella S, Rossi M, Tiranini L, Martini E. Female sexual dysfunction (FSD): Prevalence and impact on quality of life (QoL). Maturitas. 2016 Dec;94:87-91. doi: 10.1016/j.maturitas.2016.09.013. Epub 2016 Sep 28. PMID 27823751
- [Background] Kaur N, Gupta A, Sharma AK, Jain A. Survivorship issues as determinants of quality of life after breast cancer treatment: Report from a limited resource setting. Breast. 2018 Oct;41:120-126. doi: 10.1016/j.breast.2018.07.003. Epub 2018 Jul 11. PMID 30029054
- [Background] Oyarzun MFG, Castelo-Branco C. Local hormone therapy for genitourinary syndrome of menopause in breast cancer patients: is it safe? Gynecol Endocrinol. 2017 Jun;33(6):418-420. doi: 10.1080/09513590.2017.1290076. Epub 2017 Feb 21. PMID 28277141
- [Background] Lubian Lopez DM. Management of genitourinary syndrome of menopause in breast cancer survivors: An update. World J Clin Oncol. 2022 Feb 24;13(2):71-100. doi: 10.5306/wjco.v13.i2.71. PMID 35316932
- [Background] Sulaica E, Han T, Wang W, Bhat R, Trivedi MV, Niravath P. Vaginal estrogen products in hormone receptor-positive breast cancer patients on aromatase inhibitor therapy. Breast Cancer Res Treat. 2016 Jun;157(2):203-210. doi: 10.1007/s10549-016-3827-7. Epub 2016 May 13. PMID 27178335
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Pater JL. Randomized trial of letrozole following tamoxifen as extended adjuvant therapy in receptor-positive breast cancer: updated findings from NCIC CTG MA.17. J Natl Cancer Inst. 2005 Sep 7;97(17):1262-71. doi: 10.1093/jnci/dji250. PMID 16145047
- [Background] Goss PE, Ingle JN, Pritchard KI, Robert NJ, Muss H, Gralow J, Gelmon K, Whelan T, Strasser-Weippl K, Rubin S, Sturtz K, Wolff AC, Winer E, Hudis C, Stopeck A, Beck JT, Kaur JS, Whelan K, Tu D, Parulekar WR. Extending Aromatase-Inhibitor Adjuvant Therapy to 10 Years. N Engl J Med. 2016 Jul 21;375(3):209-19. doi: 10.1056/NEJMoa1604700. Epub 2016 Jun 5. PMID 27264120
- [Background] Hocke C, Diaz M, Bernard V, Frantz S, Lambert M, Mathieu C, Grellety-Cherbero M. [Genitourinary menopause syndrome. Postmenopausal women management: CNGOF and GEMVi clinical practice guidelines]. Gynecol Obstet Fertil Senol. 2021 May;49(5):394-413. doi: 10.1016/j.gofs.2021.03.025. Epub 2021 Mar 20. French. PMID 33757926
- [Background] Faubion SS, Larkin LC, Stuenkel CA, Bachmann GA, Chism LA, Kagan R, Kaunitz AM, Krychman ML, Parish SJ, Partridge AH, Pinkerton JV, Rowen TS, Shapiro M, Simon JA, Goldfarb SB, Kingsberg SA. Management of genitourinary syndrome of menopause in women with or at high risk for breast cancer: consensus recommendations from The North American Menopause Society and The International Society for the Study of Women's Sexual Health. Menopause. 2018 Jun;25(6):596-608. doi: 10.1097/GME.0000000000001121. PMID 29762200
- [Background] Loprinzi CL, Abu-Ghazaleh S, Sloan JA, vanHaelst-Pisani C, Hammer AM, Rowland KM Jr, Law M, Windschitl HE, Kaur JS, Ellison N. Phase III randomized double-blind study to evaluate the efficacy of a polycarbophil-based vaginal moisturizer in women with breast cancer. J Clin Oncol. 1997 Mar;15(3):969-73. doi: 10.1200/JCO.1997.15.3.969. PMID 9060535
- [Background] Juliato PT, Rodrigues AT, Stahlschmidt R, Juliato CR, Mazzola PG. Can polyacrylic acid treat sexual dysfunction in women with breast cancer receiving tamoxifen? Climacteric. 2017 Feb;20(1):62-66. doi: 10.1080/13697137.2016.1258396. Epub 2016 Nov 23. PMID 27876429
- [Background] Lee YK, Chung HH, Kim JW, Park NH, Song YS, Kang SB. Vaginal pH-balanced gel for the control of atrophic vaginitis among breast cancer survivors: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):922-927. doi: 10.1097/AOG.0b013e3182118790. PMID 21422866
- [Background] Advani P, Brewster AM, Baum GP, Schover LR. A pilot randomized trial to prevent sexual dysfunction in postmenopausal breast cancer survivors starting adjuvant aromatase inhibitor therapy. J Cancer Surviv. 2017 Aug;11(4):477-485. doi: 10.1007/s11764-017-0606-3. Epub 2017 Feb 22. PMID 28229275
- [Background] Edwards D, Panay N. Treating vulvovaginal atrophy/genitourinary syndrome of menopause: how important is vaginal lubricant and moisturizer composition? Climacteric. 2016 Apr;19(2):151-61. doi: 10.3109/13697137.2015.1124259. Epub 2015 Dec 26. PMID 26707589
- [Background] Palacios S, Castelo-Branco C, Currie H, Mijatovic V, Nappi RE, Simon J, Rees M. Update on management of genitourinary syndrome of menopause: A practical guide. Maturitas. 2015 Nov;82(3):308-13. doi: 10.1016/j.maturitas.2015.07.020. Epub 2015 Jul 26. PMID 26261035
- [Background] Chen J, Geng L, Song X, Li H, Giordan N, Liao Q. Evaluation of the efficacy and safety of hyaluronic acid vaginal gel to ease vaginal dryness: a multicenter, randomized, controlled, open-label, parallel-group, clinical trial. J Sex Med. 2013 Jun;10(6):1575-84. doi: 10.1111/jsm.12125. Epub 2013 Apr 9. PMID 23574713
- [Background] Ekin M, Yasar L, Savan K, Temur M, Uhri M, Gencer I, Kivanc E. The comparison of hyaluronic acid vaginal tablets with estradiol vaginal tablets in the treatment of atrophic vaginitis: a randomized controlled trial. Arch Gynecol Obstet. 2011 Mar;283(3):539-43. doi: 10.1007/s00404-010-1382-8. Epub 2010 Feb 5. PMID 20135132
- [Background] Speroff L. The LIBERATE tibolone trial in breast cancer survivors. Maturitas. 2009 May 20;63(1):1-3. doi: 10.1016/j.maturitas.2009.03.001. Epub 2009 Mar 26. No abstract available. PMID 19327923
- [Background] Holmberg L, Anderson H; HABITS steering and data monitoring committees. HABITS (hormonal replacement therapy after breast cancer--is it safe?), a randomised comparison: trial stopped. Lancet. 2004 Feb 7;363(9407):453-5. doi: 10.1016/S0140-6736(04)15493-7. PMID 14962527
- [Background] von Schoultz E, Rutqvist LE; Stockholm Breast Cancer Study Group. Menopausal hormone therapy after breast cancer: the Stockholm randomized trial. J Natl Cancer Inst. 2005 Apr 6;97(7):533-5. doi: 10.1093/jnci/dji071. PMID 15812079
- [Background] Biglia N, Bounous VE, Sgro LG, D'Alonzo M, Pecchio S, Nappi RE. Genitourinary Syndrome of Menopause in Breast Cancer Survivors: Are We Facing New and Safe Hopes? Clin Breast Cancer. 2015 Dec;15(6):413-20. doi: 10.1016/j.clbc.2015.06.005. Epub 2015 Jun 18. PMID 26198332
- [Background] Behnia-Willison F, Sarraf S, Miller J, Mohamadi B, Care AS, Lam A, Willison N, Behnia L, Salvatore S. Safety and long-term efficacy of fractional CO2 laser treatment in women suffering from genitourinary syndrome of menopause. Eur J Obstet Gynecol Reprod Biol. 2017 Jun;213:39-44. doi: 10.1016/j.ejogrb.2017.03.036. Epub 2017 Apr 2. PMID 28419911
- [Background] Maris E, Salerno J, Hedon B, Mares P. [Management of vulvovaginal atrophy: Physical therapies. Postmenopausal women management: CNGOF and GEMVi clinical practice guidelines]. Gynecol Obstet Fertil Senol. 2021 May;49(5):414-419. doi: 10.1016/j.gofs.2021.03.021. Epub 2021 Mar 20. French. PMID 33757917
- [Background] Pitsouni E, Grigoriadis T, Falagas ME, Salvatore S, Athanasiou S. Laser therapy for the genitourinary syndrome of menopause. A systematic review and meta-analysis. Maturitas. 2017 Sep;103:78-88. doi: 10.1016/j.maturitas.2017.06.029. Epub 2017 Jun 27. PMID 28778337
- [Background] Pitsouni E, Grigoriadis T, Douskos A, Kyriakidou M, Falagas ME, Athanasiou S. Efficacy of vaginal therapies alternative to vaginal estrogens on sexual function and orgasm of menopausal women: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:45-56. doi: 10.1016/j.ejogrb.2018.08.008. Epub 2018 Aug 6. PMID 30103082
- [Background] Jha S, Wyld L, Krishnaswamy PH. The Impact of Vaginal Laser Treatment for Genitourinary Syndrome of Menopause in Breast Cancer Survivors: A Systematic Review and Meta-analysis. Clin Breast Cancer. 2019 Aug;19(4):e556-e562. doi: 10.1016/j.clbc.2019.04.007. Epub 2019 Apr 19. PMID 31227415
- [Background] Cruz VL, Steiner ML, Pompei LM, Strufaldi R, Fonseca FLA, Santiago LHS, Wajsfeld T, Fernandes CE. Randomized, double-blind, placebo-controlled clinical trial for evaluating the efficacy of fractional CO2 laser compared with topical estriol in the treatment of vaginal atrophy in postmenopausal women. Menopause. 2018 Jan;25(1):21-28. doi: 10.1097/GME.0000000000000955. PMID 28763401
- [Background] Ruanphoo P, Bunyavejchevin S. Treatment for vaginal atrophy using microablative fractional CO2 laser: a randomized double-blinded sham-controlled trial. Menopause. 2020 Aug;27(8):858-863. doi: 10.1097/GME.0000000000001542. PMID 32345787
- [Background] Paraiso MFR, Ferrando CA, Sokol ER, Rardin CR, Matthews CA, Karram MM, Iglesia CB. A randomized clinical trial comparing vaginal laser therapy to vaginal estrogen therapy in women with genitourinary syndrome of menopause: The VeLVET Trial. Menopause. 2020 Jan;27(1):50-56. doi: 10.1097/GME.0000000000001416. PMID 31574047
- [Background] Filippini M, Porcari I, Ruffolo AF, Casiraghi A, Farinelli M, Uccella S, Franchi M, Candiani M, Salvatore S. CO2-Laser therapy and Genitourinary Syndrome of Menopause: A Systematic Review and Meta-Analysis. J Sex Med. 2022 Mar;19(3):452-470. doi: 10.1016/j.jsxm.2021.12.010. Epub 2022 Jan 29. PMID 35101378
- [Background] Gordon C, Gonzales S, Krychman ML. Rethinking the techno vagina: a case series of patient complications following vaginal laser treatment for atrophy. Menopause. 2019 Apr;26(4):423-427. doi: 10.1097/GME.0000000000001293. PMID 30640806
- [Background] Al-Badr A, Alkhamis WH. Laser Vaginal Tightening Complications: Report of Three Cases. Lasers Surg Med. 2019 Nov;51(9):757-759. doi: 10.1002/lsm.23110. Epub 2019 Jun 18. PMID 31215051
- [Background] FDA Warns Against Use of Energy-Based devices to perform vaginal 'rejuvenation' or vaginal cosmetic procedures: FDA Safety Communication. July 30, 2018. (Updated November 20, 2018). https://www.fda.gov/medicaldevices/ safety/alertsandnotices/ucm615013.htm. Accessed March 31, 2021.
- [Background] Forret A, Mares P, Delacroix C, Chevallier T, Potier H, Fatton B, Masia F, Ripart S, Letouzey V, de Tayrac R, Salerno J. [Photobiomodulation and vulvovaginal disorders after anticancer treatments]. Bull Cancer. 2023 Sep;110(9):883-892. doi: 10.1016/j.bulcan.2023.03.018. Epub 2023 May 12. French. PMID 37183056
- [Background] Hantash BM, Ubeid AA, Chang H, Kafi R, Renton B. Bipolar fractional radiofrequency treatment induces neoelastogenesis and neocollagenesis. Lasers Surg Med. 2009 Jan;41(1):1-9. doi: 10.1002/lsm.20731. PMID 19143021
- [Background] Coad J, Vos J, Curtis A, Krychman M. Safety and mechanisms of action supporting nonablative radiofrequency thermal therapy for vaginal introitus laxity occurring in women after childbirth: histological study in the sheep vaginal model. J Sex Med 2013;10:175.
- [Background] Vanaman Wilson MJ, Bolton J, Jones IT, Wu DC, Calame A, Goldman MP. Histologic and Clinical Changes in Vulvovaginal Tissue After Treatment With a Transcutaneous Temperature-Controlled Radiofrequency Device. Dermatol Surg. 2018 May;44(5):705-713. doi: 10.1097/DSS.0000000000001453. PMID 29701623
- [Background] Sarmento AC, Fernandes FS, Marconi C, Giraldo PC, Eleuterio-Junior J, Crispim JC, Goncalves AK. Impact of microablative fractional radiofrequency on the vaginal health, microbiota, and cellularity of postmenopausal women. Clinics (Sao Paulo). 2020;75:e1750. doi: 10.6061/clinics/2020/e1750. Epub 2020 Aug 3. PMID 32756817
- [Background] Elbiss HM, Rafaqat W, Khan KS. The effect of dynamic quadripolar radiofrequency on genitourinary atrophy and sexual satisfaction: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Oct 7;101(40):e30960. doi: 10.1097/MD.0000000000030960. PMID 36221421
- [Background] Vicariotto F, Raichi M. Technological evolution in the radiofrequency treatment of vaginal laxity and menopausal vulvo-vaginal atrophy and other genitourinary symptoms: first experiences with a novel dynamic quadripolar device. Minerva Ginecol. 2016 Jun;68(3):225-36. PMID 27206062
- [Background] Benincà G, Bosoni D, Vicariotto F, et al. Efficacy and safety of Dynamic Quadripolar RadioFrequency, a new high-tech, highsafety option for vulvar rejuvenation. Obstet Gynecol Reports. 2017;1.
- [Background] Fasola E, Bosoni D. Dynamic Quadripolar Radiofrequency: Pilot Study of a New High-Tech Strategy for Prevention and Treatment of Vulvar Atrophy. Aesthet Surg J. 2019 Apr 8;39(5):544-552. doi: 10.1093/asj/sjy180. PMID 30052757
- [Background] Leibaschoff G, Izasa PG, Cardona JL, Miklos JR, Moore RD. Transcutaneous Temperature Controlled Radiofrequency (TTCRF) for the Treatment of Menopausal Vaginal/Genitourinary Symptoms. Surg Technol Int. 2016 Oct 26;29:149-159. PMID 27608749
- [Background] Sarmento ACA, Fernandes FS, Costa APF, Medeiros KS, Crispim JC, Goncalves AK. Microablative fractional radiofrequency for the genitourinary syndrome of menopause: protocol of randomised controlled trial. BMJ Open. 2021 Jul 5;11(7):e046372. doi: 10.1136/bmjopen-2020-046372. PMID 34226218
- [Background] Vicariotto F, DE Seta F, Faoro V, Raichi M. Dynamic quadripolar radiofrequency treatment of vaginal laxity/menopausal vulvo-vaginal atrophy: 12-month efficacy and safety. Minerva Ginecol. 2017 Aug;69(4):342-349. doi: 10.23736/S0026-4784.17.04072-2. PMID 28608667
- [Background] Di Maio M, Basch E, Denis F, Fallowfield LJ, Ganz PA, Howell D, Kowalski C, Perrone F, Stover AM, Sundaresan P, Warrington L, Zhang L, Apostolidis K, Freeman-Daily J, Ripamonti CI, Santini D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. The role of patient-reported outcome measures in the continuum of cancer clinical care: ESMO Clinical Practice Guideline. Ann Oncol. 2022 Sep;33(9):878-892. doi: 10.1016/j.annonc.2022.04.007. Epub 2022 Apr 21. No abstract available. PMID 35462007
- [Background] Di Maio M, Gallo C, Leighl NB, Piccirillo MC, Daniele G, Nuzzo F, Gridelli C, Gebbia V, Ciardiello F, De Placido S, Ceribelli A, Favaretto AG, de Matteis A, Feld R, Butts C, Bryce J, Signoriello S, Morabito A, Rocco G, Perrone F. Symptomatic toxicities experienced during anticancer treatment: agreement between patient and physician reporting in three randomized trials. J Clin Oncol. 2015 Mar 10;33(8):910-5. doi: 10.1200/JCO.2014.57.9334. Epub 2015 Jan 26. PMID 25624439